CLINICAL TRIAL: NCT06897631
Title: Robot-Assisted Tai Chi for Upper Limb Rehabilitation in Post-Stroke Patients: A Randomized Controlled Trial on Motor Recovery
Brief Title: Robot-Assisted Tai Chi for Upper Limb Rehabilitation in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jing Tao (Other)
Responsible Party: Sponsor-Investigator, Jing Tao, Professor, Fujian University of Traditional Chinese Medicine
Organization: Fujian University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FujianUTCM-4
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: stroke; upper limb; robot; tai chi; motor function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai Chi-based rehabilitation robot group (Experimental)
  Interventions: Device: Robot-Assisted Tai Chi Training
- Conventional rehabilitation group (Experimental)
  Interventions: Behavioral: Conventional rehabilitation training

INTERVENTIONS:
Device: Robot-Assisted Tai Chi Training — This intervention involves robot-assisted Tai Chi training for upper limb rehabilitation, delivered in a seated position to ensure participant safety and comfort. Each 60-minute session consists of a 5-minute warm-up/preparation phase, followed by three 15-minute segmented functional training phases incorporating Tai Chi-inspired movements to target upper limb coordination, range of motion, and strength recovery, interspersed with two 5-minute rest intervals. The protocol is administered 5 times per week over 4 weeks, with robotic assistance tailored to guide functional upper limb trajectories while minimizing compensatory movements.
  Arms: Tai Chi-based rehabilitation robot group
Behavioral: Conventional rehabilitation training — This intervention follows evidence-based clinical guidelines for post-stroke upper limb rehabilitation, focusing on therapist-guided task-oriented training that integrates activities of daily living (ADL) such as table wiping and clothes hanging. Sessions emphasize progressive functional integration, with exercises adjusted weekly based on patient performance. Training is delivered in 60-minute sessions (1 session/day), 5 days per week over 4 weeks, under direct therapist supervision to ensure proper movement patterns and safety.
  Arms: Conventional rehabilitation group

SUMMARY:
This study aims to compare the effectiveness of Robot-Assisted Tai Chi Training (RATT) versus conventional rehabilitation in improving upper limb motor function post-stroke, and to explore the neuromuscular mechanisms of RATT. Participants will be randomly assigned to one of two groups:

1. Robot-Assisted Tai Chi Training group: Participants will receive guided Tai Chi arm movements with robotic assistance to enhance coordination and strength.
2. Conventional rehabilitation group: Participants will perform standard exercises (e.g., stretching, repetitive task practice).

Both groups will receive 60-minute sessions, administered 5 days a week, over 4 weeks. Researchers will measure improvements using clinical scales (e.g., Fugl-Meyer Assessment) and monitor safety.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with stroke confirmed by neuroimaging (CT/MRI).
2. Fugl-Meyer Assessment for Upper Extremity score of 8-44.
3. First-ever stroke, with unilateral hemiplegia and time since onset ≤12 months.
4. Aged 40-80 years, regardless of gender.
5. Voluntarily participated and provided written informed consent. Participants meeting all above criteria were enrolled.

Exclusion Criteria:

1. Severe cognitive impairment (Montreal Cognitive Assessment score <10).
2. Poor sitting balance (< Grade 2) or inability to maintain seated position for >60 minutes.
3. Hypertonia (modified Ashworth Scale score >2 in affected limb).
4. Significant hemiplegic shoulder pain (Visual Analogue Scale >3).
5. Severe aphasia (Boston Diagnostic Aphasia Examination score <3).
6. Severe visual impairment precluding robot-assisted upper limb training.
7. Moderate-to-severe depression (17-item Hamilton Depression Rating Scale score >17).
8. Pre-existing neuromuscular disorders, active malignancies, or uncontrolled systemic diseases (cardiac, renal, hepatic).
9. Concurrent participation in other clinical trials affecting study outcomes. Participants meeting any of the above criteria were excluded.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity Scale | 4 weeks (post-intervention)
  Score range 0-66, higher scores indicate better upper limb motor recovery.

SECONDARY OUTCOMES:
Wolf Motor Function Test | 4 weeks
  The Wolf Motor Function Test (WMFT) evaluates upper limb motor function in conditions like stroke through 15 timed functional tasks (e.g., lifting objects) and 2 strength tasks. It scores Performance Time (total seconds; lower = faster) and Functional Ability (0-5 per task, max 75; higher = better movement quality), with improved motor recovery indicated by reduced time and increased ability scores.
Shoulder Range of Motion | 4 weeks
  Shoulder active (AROM) and passive (PROM) range of motion were assessed in flexion, abduction, and rotation using a standardized protocol.
Upper Limb Muscle Strength Assessment | 4 weeks
  Muscle strength is assessed using Manual Muscle Testing (MMT) graded via the Medical Research Council (MRC) Scale (range: 0-5, where 0 = no muscle contraction and 5 = normal strength, higher scores indicate better outcomes).
Trunk Impairment Scale | 4 weeks
  The 17-item Trunk Impairment Scale (TIS) comprises three subscales: static sitting balance (3 items), dynamic sitting balance (10 items), and coordination (4 items). Each item is scored on a 2-, 3- or 4-point ordinal scale from 0 to 3, with the maximal scores for the static and dynamic sitting balance and coordination subscales that can be attained being 7, 10 and 6. The total scores for the TIS range from 0 to 23, representing the lowest to the highest level of body balancing function.
Modified Barthel Index | 4 weeks
  Score range 0-100, higher scores indicate better independence in activities of daily living.
Stroke-Specific Quality of Life Scale | 4 weeks
  Score range 49-245, higher scores indicate better health-related quality of life in stroke survivors.

OTHER OUTCOMES:
Upper Limb Muscle Synergy Patterns | 4 weeks
  Surface electromyography (sEMG) signals were collected from upper limb muscles during drinking and forward-reaching tasks. Muscle synergy patterns underlying these functional movements were extracted and analyzed using non-negative matrix factorization (NMF).
Kinematic Analysis of Upper Limb Movements During Functional Motor Tasks | 4 weeks
  Upper limb kinematic data (movement trajectories and joint angles) were acquired via the OpenCap system during drinking and forward-reaching tasks. Joint moments were subsequently estimated using inverse dynamics, and task-specific motor patterns were extracted to quantify kinematic synergies and torque profiles.
Multimodal Neuroimaging Analysis | 4 weeks
  Structural (T1-MPRAGE) and resting-state fMRI data were acquired using a 3T MRI scanner. Structural analysis assessed gray matter volume and density, cortical thickness, and surface area, while functional analysis evaluated amplitude of low-frequency fluctuations (ALFF), regional homogeneity (ReHo), functional connectivity (FC), and graph theory-based network topology metrics (global/local efficiency).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Rehabilitation Hospital Affiliated to Fujian University of Traditional Chinese Medicine, Fuzhou, Fujian
  - The Third People's Hospital Affiliated to Fujian University of Traditional Chinese Medicine, Fuzhou, Fujian

IPD SHARING:
Plan to Share IPD: No